CLINICAL TRIAL: NCT00827385
Title: Impact of Intraoperative Blood Pressure on Cognitive Performance in Patients With and Without Hypertension: a Prospective Observational Study
Brief Title: Intraoperative Blood Pressure and Cognitive Performance
Status: Completed | Type: Observational
Sponsor: Weill Medical College of Cornell University (Other)
Responsible Party: Sponsor
Other Study IDs: 0809009986
Record Dates: First submitted 2009-01-21; First posted 2009-01-22 (Estimated); Last update posted 2015-02-04 (Estimated); Status verified 2015-02

CONDITIONS: Cognitive Performance; Hypertension
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- hypertensive
- normotensive

SUMMARY:
The purpose of this study is to prospectively determine the association between incidence of neurological morbidity and minimum fractional blood pressure reached during laminectomy procedures under general anesthesia in hypertensive and normotensive subjects 40 years old and older.

ELIGIBILITY:
Inclusion Criteria:

* English as first language, or as a learned language as long as the patient is proficient
* No history of any neurological disease with the exception of patients without functional impairment who suffered a single episode of transient ischemic attack
* No history of axis I psychiatric diagnosis or drug abuse
* 40 years old or older
* Undergoing laminectomy under general anesthesia
* Must not take antihypertensive medication for purposes other than treatment of hypertension

Exclusion Criteria:

* Anyone who do not fit the inclusion criteria.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: - individuals 40 years of age and older, undergoing laminectomy under general anesthesia.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2009-01; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
post-operative cognitive performance | 1

CONTACTS AND LOCATIONS:
Locations (1):
- NewYork-Presbyterian Hospital-Weill Cornell Medical College, New York, New York, United States